CLINICAL TRIAL: NCT04206644
Title: Systemic Sclerosis and Jak Inhibitors : Emphasis on Macrophages
Acronym: SCLERO JAK
Status: Active, not recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30043_SCLERO JAK
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; macrophage; ruxolitinib
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Systemic sclerosis patients: SSc patients according to the ACR/EULAR 2013 classification criteria
  Interventions: Other: biological analysis
- Healthy donors: HD healthy donors from EFS (Etablissement Français du sang)
  Interventions: Other: biological analysis
- LUPUS Patiets: Lupus patients according to the ACR 2019 classification criteria

INTERVENTIONS:
Other: biological analysis — biological analysis of the Concentration of CCL18
  Groups: Healthy donors; Systemic sclerosis patients

SUMMARY:
The Sclero-JAK project aims to assess the impact of a JAK1/2 inhibitor (ruxolitinib) on activation states of monocytes-derived macrophages (MDM) from systemic sclerosis (SSc) patients

DETAILED DESCRIPTION:
Systemic sclerosis is a fibrotic and inflammatory chronic autoimmune disorder with no disease modifiying drug available to date. JAK inhibitors may represent a relevant therapeutic candidate for this disease;

The primary objective of this study is to characterize the impact of Ruxolitinib (a JAK ½ inhibitor) on the prof-fibrotic properties of MDM from SSc patients in vitro.

The primary outcome will be the concentration of CCL18 evaluate by ELISA in the condition media of MDM from SSc patients pre treated or not in vitro by ruxolitinib.

The secondary objectives :

1. To characterize the impact of ruxolitinib on other pro-inflammatory or pro-fibrotic cytokines
2. To characterize the impact of ruxolitinib on membrane expression of macrophagic polarization markers of MDM from SSc patients
3. To evaluate the impact of ruxolitinib on the phenotype of MDM from healthy donors exposed in vitro to the serum of SSc patients.
4. To determine the variability of the effects of ruxolitinib on MDM of SSc patients depending on key clinical characteristics (diffuse versus limited SSc, patients with or without Interstitial Lung disease ILD)

The secondary outcomes :

1. ELISA of the following cytokine evaluated in the condition media of SSc MDM pre-treated or not with ruxolitinib : PDGFbb, IL-6, CXCL10, CXCL4
2. Membrane expression (flow cytometry) of the following markers expressed by SSc MDM pre-treated or not with ruxoltinib : CD204, CD206, CD163, CD86, CMHII, TLR4.
3. Evaluation of the same cytokines and membrane markers in MDM from HD exposed to serum media of SSc patients.
4. Variation of the effect of ruxolitinib on the primary outcome (CCL18 secreted in the condition media of MDM from SSc patients) in sub groups depending on the following characteristics :

   * Auto antibodies (anticentromere, antitopoisomerase, anti RNA polymerase III or none)
   * modified Rodnan skin score
   * Digital ulcers (current or past)
   * Pulmonary involvement (Interstitial Lung disease on CT scan)
   * Heart involvement (Pulmonary arterial hypertension on echocardiography)

ELIGIBILITY:
Inclusion Criteria:

* patients with systemic sclerosis according to the ACR/EULAR 2013 classification criteria for systemic sclerosis or Patients with systemic lupus according to the ACR2019 classification criteria for systemic lupus
* with informed consent for participation to the study

Exclusion Criteria:

* patients unable to consent
* patients with anemia inferior to 7g/dL

Ages: 18 Years to 18 Years | Sex: All
Age Groups: Adult
Study Population: patients with systemic sclerosis according to the ACR/EULAR 2013 classification criteria for systemic sclerosis
  or Lupus patients according to the ACR 2019 classification criteria
  or healthy donors
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2027-02-13 (Estimated)

PRIMARY OUTCOMES:
Concentration of CCL18 in the condition media of MDM from SSc patients | through study completion, an average of 4 year
  at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Patrick JEGO, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France